CLINICAL TRIAL: NCT03744091
Title: An Open Label ,Phase I, 2-way Crossover Study Evaluating the Pharmacokinetics of Prana P1 THC Activated Capsules
Brief Title: Evaluation of the Pharmacokinetics of Prana P1 Capsules
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of The West Indies (Other)
Responsible Party: Principal Investigator, Shelly Rosemarie McFarlane, Coordinating Investigator, The University of The West Indies
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PR0PK1
Record Dates: First submitted 2018-08-01; First posted 2018-11-16 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Healthy
Keywords: cannabis
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either 10 mg or 20mg arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 mg P1 (Active Comparator): 10 mg of P1 will be administered and compared with an active dose of 20 mg P1 on crossover
  Interventions: Drug: P1
- 20 mg P1 (Active Comparator): 20 mg of P1 will be administered and compared with an active dose of 10 mg P1 on crossover
  Interventions: Drug: P1

INTERVENTIONS:
Drug: P1 — 10 mg or 20 mg of THC:THCa
  Other Names: THC:THCa (delta 9-tetrahydrocannabinol ); Prana P1

SUMMARY:
This is a single dose clinical trial to assess the Pharmacokinetics of two (2) dosages; 10 mg and 20mg of THC: THCa of Prana P1 bionutrients in healthy volunteers.

DETAILED DESCRIPTION:
Single oral dose, (10 mg Prana P1 or 20 mg Prana P1) in each period with a washout of 30 days between doses. Patents will be randomly assigned dose for the first round of the study after a thirty-day washout, patient will return to the study site and receive cross over dose.

Metabolites to be Measured:

1. THC
2. 11-OH-THC [primary secondary metabolite of THC, psychoactive]
3. THC-COOH [inactive metabolite]

The following parameters for THC, 11-OH-THC, and THC-COOH will be assessed: AUC0-t, AUC0-inf, Cmax, AUCt/inf, Tmax.

Safety will be monitored and assessed through adverse events reports, 12-lead ECG, vital signs and laboratory parameters. Each participant will undergo a psychometric evaluation using the CHAT assessment tool.

ELIGIBILITY:
Inclusion Criteria:

* Males between 18 and 55 years.
* Body weight with a Body Mass Index (BMI) range of 18.5 to 27.0 [or weight within 15% of ideal weight for participant's height and frame
* Healthy, with normal findings in the physical examination and vital signs (BP between 100-140/60-90 mmHg, Heart rate (HR) between 60 to 90 beats/min, respiration between 12 to 24 breaths/min) and no clinically-significant findings in a 12-lead ECG.
* No clinical laboratory values outside of the laboratory normal reference range, unless the investigator determines them to be not clinically significant.
* Negative for hepatitis B surface antigen, hepatitis C antibody, HIV --Willing and able to communicate well with the investigator and clinic staff, comply with the study procedure and schedule, and provide written informed consent.
* Able to understand the requirements of the study and sign Informed Consent.

Exclusion Criteria:

* Current major Axis I psychiatric disorder for which the participant is currently receiving treatment or which would make study compliance an issue.
* Any condition or therapy that, in the opinion of the investigator, may be significantly worsened by the exposure to marijuana.
* Acute disease at the time of enrolment (i.e., presence of a moderate or severe illness or infection with or without a fever).
* Febrile illness (oral temperature >37.6° C at the time of drug administration).
* Unstable chronic illnesses.
* Chronic liver, renal or inflammatory bowel disease or collagen vascular disease.
* Clinically significant elevation of Alanine transaminase(ALT) and/or Aspartate transaminase (AST).
* Active neurological disorder.
* Clinically significant uncontrolled illness or clinically significant surgery within 4 weeks prior to administration of study drug.
* Cancer within the previous 5 years, other than squamous cell or basal cell carcinoma of the skin.
* Difficulty to swallow study medication.
* Smoking more than 25 cigarettes per day.
* History of any clinical laboratory abnormality deemed significant by the Principal Investigator.
* History of serious adverse reaction or hypersensitivity to any drug.
* Bleeding tendency resulting from disease or medication rendering blood collection or the injection itself unsafe (use of antiplatelet agents is allowed).
* Coagulation disorders or receiving anticoagulant therapy.
* Inability to tolerate abstinence from caffeine for 24 hours prior to and during the study treatment phase.
* Consumption of alcohol within 24 hours prior to dosing and during the treatment phase.
* History of significant alcohol or drug abuse within one year prior to the screening visit
* Chronic use (i.e., ≥3 days per week) of marijuana based products within 3 months prior to the screening visit.
* Use of hard recreational drugs (such as cocaine, phencyclidine [PCP] and crack) within one year prior to the screening visit.
* Donation of plasma (500 mL) within 7 days prior to drug administration
* Any known or suspected allergy to any constituent of marijuana.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the Principal Investigator or Sub-Investigators, contraindicates the participant 's participation in this study.
* Use of any investigational or non-registered drug or participation in an investigational study within 30 days prior to administration of study drug.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-08-23 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration( Cmax) of following a single dose of 10 mg Prana 1 | At time points, 0, 0.5hr, 1hr, 2 hr, 3hr, 4 hr, 5hr, 6hr, 8hr, 10hr, 12 hr, 24hrs, 32hrs , 48 hrs
  Maximum plasma concentration of Prana P1 following a single dose of 10 mg of Prana P1
  1. Pk endpoints of delta 9-tetrahydrocannabinol (THC) (0-24 hours post-dose) (Cmax) of THC.
     Pk endpoints of THC(0-48 hours post-dose)
  2. PK endpoints of the analyte 11-hydroxy-delta 9-tetrahydrocannabinol (T- 0-24 hours post-dose) Mean Cmax of 11-OH-THC. Mean AUC(0-t)) of 11-OH-THC.
  3. PK endpoints of the analyte 11-carboxy-delta 9-tetrahydrocannabinol (Time: 0-24 hours post-dose) Mean Cmax of 11-COOH-THC.
Peak Plasma Concentration( Cmax) of following a single dose of 20 mg Prana 1 | At time points, 0, 0.5hr, 1hr, 2 hr, 3hr, 4 hr, 5hr, 6hr, 8hr, 10hr, 12 hr, 24hrs, 32hrs , 48 hrs
  Maximum plasma concentration of Prana P1 following a single dose of 20 mg of Prana P1
  1. Pk endpoints of delta 9-tetrahydrocannabinol (THC) (0-24 hours post-dose) (Cmax) of THC.
     Pk endpoints of THC(0-48 hours post-dose)
  2. PK endpoints of the analyte 11-hydroxy-delta 9-tetrahydrocannabinol (T- 0-24 hours post-dose) Mean Cmax of 11-OH-THC. Mean AUC(0-t)) of 11-OH-THC.
  3. PK endpoints of the analyte 11-carboxy-delta 9-tetrahydrocannabinol (Time: 0-24 hours post-dose) Mean Cmax of 11-COOH-THC.

SECONDARY OUTCOMES:
Number of participants with treatment related adverse events as assessed by CTCAE v 5.0 | up to 30 days post dose
  Number of participants who experience at least one adverse event during the treatment phase relative to the pre-treatment baseline, is presented.
  The number of participants with clinically significant changes in laboratory test parameters, relative to pre-treatment baseline. (Time Frame: screening to follow-up 30 days) 5. The number of participants with a clinically significant change in vital signs, relative to pre-treatment baseline. From screening to follow-up of 30 days) 6.The number of participants with clinically significant changes in indices of the CHAT assessment tool.
Number of participants who discontinue treatment due to side effects | up to 30 days
  Number of participants who discontinue study drug due to adverse events during treatment .

CONTACTS AND LOCATIONS:
Overall Officials: Marvin Reid, MBBS, Principal Investigator — Caribbean Institute for Health Research, University of the West Indies
Locations (1):
- Tropical Metabolism Research Unit, Caribbean Institute for Health Reserach, University of the West Indies, Mona, Kingston, Jamaica

IPD SHARING:
Plan to Share IPD: No